CLINICAL TRIAL: NCT02212626
Title: Prospective, Non-randomized Multi-center, Controlled Physician-initiated Trial: Rotarex Belgium In-stent Occlusion
Acronym: ROBINSON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-130326
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

ARMS (1):
- Rotarex (Experimental): After assessment of the lesion by angiography the occlusion is intraluminally crossed with the wire according to physician's discretion. The device is introduced and the catheter is activated while its tip is still proximal to the occlusion to allow lubrication of the spiral inside the catheter with the aspirated blood. The catheter is advanced into the occlusion with occasional retraction into the already recanalized lumen. Care must be taken to achieve sufficient cooling of the catheter tip and evacuation of the debris to get an appropriate blood flow along the catheter. In order to minimize peripheral embolization of clot the distal end of the occlusion should not be passed too fast before all loose material has been sucked back into the catheter. Several passages of the occlusion may be needed to clean out all wall-adherent thrombotic material. If residual underlying stenosis of >30% persist further endovascular treatment can be performed according to the physician's discretion.
  Interventions: Device: Rotarex S

INTERVENTIONS:
Device: Rotarex S

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of recanalization of acute and subacute femoropopliteal stent occlusions with the Rotarex S catheter (Straub Medical)

DETAILED DESCRIPTION:
The treatment of acute and subacute thromboembolic and local thrombotic ischemic lesions of the ilaco-popliteal segments in the lower extremities has undergone considerable changes over recent years. The standard modality of surgical thrombectomy with the Fogarty balloon catheter technique for acute arterial occlusions has been replaced by percutaneous catheter techniques, i.e. percutaneous aspiration thrombectomy (PAT) for thrombus aspiration. Alternatively, catheter-directed pharmacologic thrombolytic therapy with or without additional catheter aspiration is used, particularly if the occlusion is already a few days or weeks old. These techniques obtain the best results in acute occlusions of less than 2 weeks' duration.

Both techniques have limitations such as the application of fibrinolytic substances and technical, impossibility of rapid and complete thrombus extraction. Therefore various mechanical devices have been introduced which involve maceration or fragmentation and removal of thrombus. The two categories of devices for mechanical thrombectomy (MT) are: (1) rotational recirculation devices which work by the vortex principle, such as the Amplatz thrombectomy catheter (ATD, Microvena, White Bear Lake, MN) or the Arrow-Trerotola PTD (Arrow International, Reading, PA); and (2) hydrodynamic (rheolytic) recirculation devices which operate on the principle of the Venturi effect, such as the Hydrolyser (Cordis, Johnson and Johnson, Miami, FL), Oasis (Boston Scientific, Galway, Ireland), and the Angiojet (RTC; Possis Medical, Minneapolis, MN) [5-10]. These devices are not suited for subacute occlusions of more than 7-14 days' duration. Recently, a new rotational mechanical thrombectomy catheter, the Straub Rotarex / Aspirex (Straub Medical, 7323 Wangs, Switzerland) has been introduced. This device combines the two essential effects of mechanical clot fragmentation and removal of the fragmented clot material from the vessel by negative pressure. Two studies using the Rotarex system with 38, resp. 98 patients showed a primary patency rate of 62%, resp. 54% at 6 months and described the Rotarex / Aspirex systems as an efficient and quick technique for revascularization of acute femoropopliteal de novo occlusions. A more recent publication dating from 2011 reports results from using Rotarex® catheters for treatment of in-stent reocclusions of femoropopliteal arteries. In 78 patients, the restenosis rate was calculated as 18.4% after 12 months.

The purpose of this Belgian multi-center study is to follow-up patients after recanalization with the Rotarex®S catheter system (Straub Medical) for acute and subacute femoropopliteal stent occlusions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life-expectancy of at least 6 months
* Symptomatic acute or subacute stent occlusion in the femoropopliteal artery
* Target vessel diameter ≥ 3 mm and ≤ 8 mm
* Patient is candidate for thrombolytic or anticoagulation medication
* Patient is able and willing to comply with study follow-up requirements

Exclusion Criteria:

* No patent artery until the foot
* Inability of crossing lesion with guidewire
* Known active infection at the time of intervention
* Untreated flow-limiting inflow lesions
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrolment
* Aneurysm in the target vessel
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancy, dementia, etc) or other medical condition that would preclude compliance with the study protocol
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Septicemia or bacteremia
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Patient with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Currently participating in another clinical research trial
* The patient must be excluded in case any of the following contraindications as listed in the IFU is present:

Rotarex®S catheters must not be used in case of:

* Patient not suitable for thrombectomy
* Target vessel belonging to the vessels of the cardiopulmonary, coronary or cerebral circulations
* Use inside or via undersized or oversized vessel diameters
* Impossibility to pass the lesion completely with the guidewire
* Subintimal position of the guidewire - even if only in short segments
* Use in stents or stent grafts if the guidewire has become threaded at any point in the wire mesh of stent or stent graft or the lining of the stent graft
* The introducer sheath, the guide catheter, the guidewire or the Rotarex®S catheter sustaining any damage, especially kinking
* Target lesions situated in the fracture areas of broken stents
* Known or suspected allergy to any of the components of the system or to a medicinal product to be administered in connection with the planned procedure
* Persistent vasospasm
* Imaging by Magnetic Resonance Imaging (MRI)
* Use of a defibrillator on the patient
* Use of electrosurgery on the patient
* Veterinary purposes
* Patients with hemodynamic instability or shock
* Patients with severe coagulatory disorders
* Situations where an embolism potentially triggered by the use of the catheter may have a very harmful effect on the patient
* Use inside or via narrow vessel radii or in tortuous vessel courses (radius of curvature < 2cm)
* Target lesion in severely calcified vessel segments
* Target lesion in aneurysmatically altered vessel segments
* Known or suspected infection, especially of the puncture site or the vessel segment being treated
* Known, unhealed pre-existing mechanical damage to the vessel wall, especially caused by surgical procedures or interventional complications
* Impossibility to achieve sufficient anticoagulation and platelet aggregation inhibition

  * Patient is pregnant or nursing a child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Technical success of the Rotarex device | 1 day post-op
  Defined as removal of all thrombotic material, documented by angiography pre- and post-procedure: residual stenosis of the lesion <30%.
Absence of procedure related complications | 1 day post-op
  Embolization, amputation, perforation or hemorrhage.

SECONDARY OUTCOMES:
Primary patency at 6 month follow-up | 6 months
  Defined as absence of restenosis (≥50% stenosis) or occlusion within the originally treated lesion based on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without prior TLR are defined as being primary patent at the 6-month follow-up.
Target Lesion Revascularization (TLR) | 1 and 6 months
  Defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the treated lesion edge.
Clinical success | 1 and 6 months
  Defined as an improvement of Rutherford classification at 6 month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Serious Adverse Events | up to 6 months
  Defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - OLV Hospital, Aalst
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - UZA, Edegem
  - RZ Heilig Hart Hospital, Tienen